CLINICAL TRIAL: NCT00362167
Title: Evaluation and Treatment of Pain (Training Protocol)
Brief Title: Pain Evaluation and Treatment
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010092; 01-D-0092
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-12-13

CONDITIONS: Pain
Keywords: Clinical Experience; Educational Training; Pain Syndromes; Analgesia; Pain Medicine; Therapy; Neuropathic; Chronic Pain; Acute Pain; Analgesics; Medication; Evaluation
MeSH Terms: conditions — Pain; Somatoform Disorders; Agnosia; Chronic Pain; Acute Pain

SUMMARY:
This study offers evaluation and treatment for patients with a spectrum of acute and chronic pain syndromes. The protocol is not designed to test new treatments; rather, patients will receive current standard of care treatments. The purposes of the study are: 1) to allow physicians in NIDCR's Pain and Neurosensory Mechanisms Branch to gain more knowledge about treating acute and chronic pain and possibly identify new avenues of research in this area; and 2) to establish a pool of patients who may be eligible for new studies as they are developed. (Participants in this protocol will not be required to join a new study; the decision will be voluntary.)

Patients 12 years of age and older with an acute or chronic pain syndrome may be eligible for this study. Women of childbearing potential and women who are pregnant or breastfeeding will not be enrolled in this study, drugs may have unknown or untoward side effects on the baby.

Participants will provide a medical history, as well as occupational and social information. They will have a standard neurological examination, including a test of cognitive (thinking) abilities, muscular function, reflexes and sensory examination. The latter involves testing with a pin placed on the surface of the skin. Participants will also have routine blood tests and will fill out questionnaires on their daily functioning and psychological well being. Additional procedures may include magnetic resonance imaging (MRI) scans and possible referral to a psychiatrist for evaluation of depression or emotional difficulties.

Participants will be treated according to their individual pain problem. Treatments may include medicines, exercises, physical therapy, nerve blocks and dietary changes. Medicines given in this study are commonly used by doctors to treat pain, but for many, there is little research to back up their use. This study will provide information on the effectiveness of these treatments. Participants will keep a daily log in which they rate their pain, record any procedures they undergo outside the study, such as injections and exercises, and record medication side effects.

Participation in the study will end based on the researcher's assessment of the patient's response to treatment. The study doctor will provide the patient's referring doctor a report of medications or other treatments used in the study. At the last visit, patients will fill out the same questionnaires they filled out during the first visit.

DETAILED DESCRIPTION:
The function of this protocol is to allow the clinic pain research fellows to gain additional knowledge in the management of acute and chronic pain. Patients enrolled in this protocol will be evaluated and treated according to available procedures and therapeutic modalities used in clinical practice. The evaluation and treatment of these patients may lead to ideas for future protocols.

By allowing for the care of persons with a spectrum of pain syndromes, this protocol will be valuable for the training of the pain fellow as well. The pain group at the NIDCR is free to choose those diseases that interest them.

Patients in this patient evaluation and treatment protocol will be evaluated for potential eligibility in any of the new clinical studies of the Pain and Neurosensory Mechanisms branch of the NIDCR as they are developed. If eligible, patients may be asked to participate in the new protocol. However they will not be required to enter any new protocol and their decision to participate will be entirely voluntary.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients of 4 years of age and older, both genders, and all racial/ethnic groups with acute or chronic pain that will help the Branch fulfill its objectives.

Women of childbearing potential, or who are pregnant or lactating, will only undergo tests and procedures, and/or receive medications for which data exists proving minimal risk to the fetus. The diagnostic tests will only include medically-indicated radiation exposure.

Referral is needed from the patients' physician or dentist.

EXCLUSION CRITERIA:

Patients with significant cognitive impairment.

Pregnancy or lactation, if this status precludes proposed diagnostic procedures or therapies.

Patients with serious organ system dysfunction (e.g. heart failure, ischemic heart disease).

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2001-02-15; Study Completion 2006-12-13

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States